CLINICAL TRIAL: NCT00264082
Title: "Tartrate-Resistant Acid Phosphatase as a Bone Resorption Marker in Stage IV Breast Cancer Patients With Bone Metastasis During Zometa Treatment: A Pilot Study"
Brief Title: Assessment of Tartrate-Resistant Acid Phosphatase (TRAP) as a Bone Resorption Marker in Stage IV Breast Cancer Patients With Bone Metastasis
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 419.04
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Other

INTERVENTIONS:
Drug: Zometa(drug)

SUMMARY:
The purpose of this research study is to evaluate the usefulness of the TRAP protein as (1) an early indicator of bone destruction and (2) a tool for assessing the effect of Zometa® in treating symptoms of bone metastases due to breast cancer. Tartrate-resistant acid phosphatase (TRAP) is a protein released into the blood stream as a result of bone destruction caused by metastasis of breast cancer to the bone. Bone destruction causes pain and bone fractures. This study will measure TRAP levels in serum taken from breast cancer patients to see if TRAP levels will be able to predict the effect of Zometa® treatment on bone destruction, pain and bone fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic documentation of breast cancer.
2. Stage IV Breast Cancer Patients with bone metastasis for whom Zometa treatment will be initiated.
3. Age > 18
4. Written informed consent prior to study entry
5. Patients may be currently receiving hormone therapy, chemotherapy and/or radiation therapy to the primary tumor.
6. Life expectancy of at least 6 months.
7. We will include patients who have had previous or current radiation therapy to breast

Exclusion Criteria:

1. Concurrent malignancy with a second primary
2. Stage I, Stage II and Stage III
3. ECOG Performance Status 3 or 4.
4. Renal Failure - serum creatinine >2.O mg/dL at screening
5. AST or ALT > ULN X 3. at screening
6. Bilirubin > 3.0 mg/dL at screening
7. Pregnant women
8. Prior or current bisphosphonate therapy
9. Any skeletal related event due to malignancy prior to study enrollment.
10. Patients with osteoporotic fractures prior to study enrollment.
11. Allergy to bisphosphonates
12. Any radiation therapy for the treatment of bone metastases <4 weeks prior to study start.
13. Any chronic medical condition which would preclude performance or adherence to protocol requirements
14. Inability to provide informed consent

    -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-09; Primary Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leela Bhupalam, MD, Principal Investigator — University of Louisville, James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, 529 S. Jackson St., Louisville, Kentucky, United States

REFERENCES:
- See also: Related Info — http://browncancercenter.org